CLINICAL TRIAL: NCT00895011
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Study of the Safety and Efficacy of Avanafil in the Treatment of Erectile Dysfunction Following Bilateral Nerve-Sparing Radical Prostatectomy
Brief Title: Research Evaluating an Investigational Medication for Erectile Dysfunction - Post-Prostatectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TA-303; NCT01171001 (obsolete NCT alias)
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; E.D.
MeSH Terms: conditions — Erectile Dysfunction | interventions — avanafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Avanafil 100 mg (Experimental)
  Interventions: Drug: Avanafil
- Avanafil 200 mg (Experimental)
  Interventions: Drug: Avanafil

INTERVENTIONS:
Drug: Placebo — One dose 30 minutes prior to initiation of sexual activity
  Arms: Placebo
Drug: Avanafil — One dose 30 minutes prior to initiation of sexual activity
  Other Names: TA-1790; Stendra
  Arms: Avanafil 100 mg
Drug: Avanafil — One dose 30 minutes prior to initiation of sexual activity
  Other Names: TA-1790; Stendra
  Arms: Avanafil 200 mg

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of two doses of avanafil in the treatment of adult males for erectile dysfunction following bilateral nerve-sparing radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult males ≥ 18 years and ≤ 70 years;
* Have a history of erectile dysfunction of at least 6 months duration following bilateral nerve-sparing retropubic radical prostatectomy;
* Have a PSA level consistent with the absence of prostate cancer;
* Have a history of sexual potency prior to radical prostatectomy without requiring medical therapy;
* Be in a monogamous, heterosexual relationship with their current partner for at least 3 months;
* Provide written informed consent;
* Agree to make at least 4 attempts at intercourse per month;
* Agree not to use any other treatments for erectile dysfunction;
* Be willing and able to comply with all study requirements (including scheduled study visits, treatment plans, laboratory tests and other study procedures).

Exclusion Criteria

* Allergy or hypersensitivity to PDE5 inhibitors or any of the components of these drug products;
* History of dose-limiting AEs during prior treatment with a PDE5 inhibitor or discontinued use of a PDE5 inhibitor due to lack of efficacy at the highest tolerated dose;
* Concomitant use of one or more of the following medications:

  * Any nitrate, trazodone, itraconazole, ketoconazole, erythromycin, or cimetidine;
  * Other prescription or OTC drugs that are known to interfere with metabolism by the CYP 3A4 enzyme;
  * If receiving hormone replacement therapy (including thyroid supplementation), dose that has not been stable for at least 3 months;
  * If treated with an alpha blocker, dose that has not been stable for at least 14 days;
* Erectile dysfunction as a consequence of advanced neurologic disease, spinal cord injury, or diabetes;
* History of severe erectile dysfunction requiring medical therapy prior to bilateral nerve-sparing radical prostatectomy;
* History of previous pelvic surgery, brachytherapy, or cryotherapy of the prostate;
* Sexual partner who is under 18 years of age, pregnant, intends to become pregnant during the course of the study, is breastfeeding, has dyspareunia or other gynecologic conditions or other major medical conditions that would interfere with sexual activity or would have difficulty complying with study requirements;
* Uncontrolled hypertension;
* Hypotension;
* Orthostatic hypotension;
* Myocardial infarction, stroke, life-threatening arrhythmia or coronary revascularization within the past 6 months;
* Unstable angina, angina with sexual intercourse, or congestive heart failure > NYHA Class II;
* History or ECG evidence of any high-risk arrhythmia or clinically significant ECG;
* Hypertrophic, obstructive, or other clinically significant cardiomyopathy, moderate or severe cardiac valvular disease;
* Type 1 or type 2 diabetes, history of use of any antidiabetic medication;
* Clinically evident penile lesions, abrasions, anatomical deformities such as penile fibrosis, Peyronie's disease, penile implants, urinary tract or bladder infection, or sexually transmissible disease that the investigator deems to be clinically significant;
* Condition(s) predisposing to priapism, such as sickle cell disease , multiple myeloma, or leukemia;
* Any malignancy other than carcinoma of the prostate (except basal cell carcinoma or squamous cell carcinoma of the skin);
* Prior use of, or likely to require radiotherapy, chemotherapy, androgen deprivation therapy, cryotherapy, non-nerve-sparing surgery, and/or bladder or penile surgery during the study;
* Evidence of significant hepatic impairment;
* On dialysis, or history of renal transplantation;
* Untreated hypogonadism or low serum total testosterone;
* Abnormal laboratory value(s) judged to be clinically significant by the investigator;
* Positive STD screen (syphilis, gonorrhea, or chlamydia);
* Positive for HIV, HCV Ab, or HBsAg at screening;
* History or current drug, alcohol, or substance abuse;
* Positive urine drug screen;
* Positive breath alcohol test;
* Retinitis pigmentosa or nonarteritic anterior ischemic optic neuropathy;
* Use of any treatment or device for treatment of erectile dysfunction;
* Use of any other investigational medication or device for any indication within 30 days prior to enrollment or at any time during this study;
* Previous participation in any other investigational study of avanafil;
* Any history of bipolar disorder or psychosis, greater than one lifetime episode of major depression, current depression of moderate or greater severity or antidepressant use that has not been stable for at least 3 months;
* Involvement in the planning and conduct of the study on the part of subject or partner;
* Evidence of any clinically significant medical, psychiatric, social or other condition by history, physical examination or laboratory studies that, in the opinion of the investigator, would contraindicate the administration of study medications, affect compliance, interfere with study evaluations, limit study participation, contraindicate sexual activity or confound the interpretation of study results.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mulhall, MD, Study Director — Memorial Sloan Kettering Cancer Center
Locations (45):
- United States (45):
  - Research Site, Phoenix, Arizona
  - Research Site, Laguna Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, Aurora, Colorado
  - Research Site, Englewood, Colorado
  - Research Site, Parker, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Trinity, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Brighton, Massachusetts
  - Research Site, Burlington, Massachusetts
  - Research Site, Jamaica Plain, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Hackensack, New Jersey
  - Research Site, Lawrenceville, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Garden City, New York
  - Research Site, Great Neck, New York
  - Research Site, New York, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Bala-Cynwyd, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Temple, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Richmond, Virginia

REFERENCES:
- [Derived] Mulhall JP, Burnett AL, Wang R, McVary KT, Moul JW, Bowden CH, DiDonato K, Shih W, Day WW. A phase 3, placebo controlled study of the safety and efficacy of avanafil for the treatment of erectile dysfunction after nerve sparing radical prostatectomy. J Urol. 2013 Jun;189(6):2229-36. doi: 10.1016/j.juro.2012.11.177. Epub 2012 Dec 3. PMID 23219537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred at US investigative sites between April 2009 and December 2010.
Pre-assignment Details: Subjects meeting the initial eligibility criteria completed a 4-week non-treatment run-in period during which information on each attempt at intercourse was recorded. At the end of the run-in, subjects meeting the randomization criteria were eligible for assignment to one of the treatment groups.
Groups:
- Placebo: placebo 30 minutes orally prior to initiation of sexual activity
- Avanafil 100 mg: avanafil 100 mg 30 minutes orally prior to initiation of sexual activity
- Avanafil 200 mg: avanafil 200 mg 30 minutes orally prior to initiation of sexual activity
Period: Overall Study
Arm/Group | Placebo | Avanafil 100 mg | Avanafil 200 mg
Started | 100 | 99 | 99
Completed | 76 | 85 | 91
Not Completed | 24 | 14 | 8
Not completed — Withdrawal by Subject | 14 | 7 | 2
Not completed — Lost to Follow-up | 5 | 4 | 1
Not completed — Protocol Violation | 3 | 1 | 3
Not completed — Adverse Event | 1 | 2 | 2
Not completed — schedule conflict | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Avanafil 100 mg | Avanafil 200 mg | Total
Number analyzed (Participants) | 100 | 99 | 99 | 298
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 85 | 81 | 84 | 250
  >=65 years | 15 | 18 | 15 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 58.6 (5.87) | 58.9 (5.88) | 57.7 (6.60) | 58.4 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 100 | 99 | 99 | 298
Region of Enrollment [Number; unit: participants]
  United States | 100 | 99 | 99 | 298

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Sexual Attempts in Which Subjects Are Able to Maintain an Erection of Sufficient Duration to Have Successful Intercourse
Description: Data presented as mean change from baseline in the percentage of Yes responses to Sexual Encounter Profile (SEP) diary question 3 "Did your erection last long enough for you to have successful intercourse?"
Time Frame: Baseline, Week 12
Population: Number of participants analyzed represents the Intent-to-Treat population.
Measure: Least Squares Mean (Standard Error); unit: percentage of sexual attempts
Groups:
- Placebo: placeb 30 minutes orally prior to initiation of sexual activity
Arm/Group | Placebo | Avanafil 100 mg | Avanafil 200 mg
Number analyzed (Participants) | 96 | 94 | 96
percentage of sexual attempts | 13.9 (3.42) | 28.0 (3.54) | 29.4 (3.33)

2. Primary Outcome: The Change in Percentage of Sexual Attempts in Which Subjects Are Able to Insert the Penis Into the Partner's Vagina
Description: Data presented as mean change from baseline in the percentage of Yes responses to Sexual Encounter Profile (SEP) diary question 2 "Were you able to insert your penis into your partner's vagina?"
Time Frame: Baseline, Week 12
Population: Number of participants analyzed represents the Intent-to-Treat population.
Measure: Least Squares Mean (Standard Deviation); unit: Percentage of Sexual Attempts
Arm/Group | Placebo | Avanafil 100 mg | Avanafil 200 mg
Number analyzed (Participants) | 96 | 94 | 96
Percentage of Sexual Attempts | 7.5 (3.68) | 22.3 (3.66) | 27.7 (3.48)

3. Primary Outcome: Change in International Index of Erectile Function - Erectile Function Domain (IIEF-EF) Score
Description: Questionnaire assesses subject's evaluation of erectile function over the previous 4-week period. Total scores from questions 1-5 & 15 range from 1 to 30. A higher score indicates better erectile function.
Time Frame: Baseline, End of Treatment (up to 12 weeks)
Population: Number of participants analyzed represents the Intent-to-Treat population. For dropouts or missing data, the last observation carried forward convention was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Avanafil 100 mg | Avanafil 200 mg
Number analyzed (Participants) | 95 | 94 | 96
scores on a scale | 1.2 (1.16) | 4.7 (1.18) | 6.2 (1.11)

ADVERSE EVENTS:
Time Frame: AE reporting began when the subject provided written informed consent and extended until 28 calendar days after the last dose of the investigational product was administered, or until the subject was discontinued from the study, whichever was later.
Description: A treatment-emergent adverse event (TEAE) is an adverse event occurring on or after the first dose of study medication, or on or after the first dispensed date if missing, and prior to the last visit.
Arm/Group | Placebo | Avanafil 100 mg | Avanafil 200 mg
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/99 | 0/99
Other Adverse Events (participants affected / at risk) | 1/100 | 16/99 | 27/99
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=100) | Avanafil 100 mg (N=99) | Avanafil 200 mg (N=99)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 1 (1) | 8 (19) | 12 (35)
Flushing (Vascular disorders) | 0 (0) | 5 (30) | 10 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's written notification that publication of results is no longer planned or 12 months after termination of the study at all sites, Institution & PI may publish, upon written approval from Sponsor, results of the Study. Sponsor will be given the opportunity to review any proposed publication at least 60 days prior to submission for publication or disclosure. Upon Sponsor's written request, Institution and PI shall not publish or disclose information related to the Study.